CLINICAL TRIAL: NCT00702676
Title: A Double-blind, Double-dummy, Randomized, Crossover Study to Compare the Tolerability of Quetiapine Fumarate Immediate Release (SEROQUEL®) With Quetiapine Fumarate Extended Release (SEROQUEL XR®) During Initial Dose Escalation in Healthy Volunteers
Brief Title: Quetiapine Fumarate Immediate Release (IR) Versus Extended Release (XR) Dose Escalation Comparison
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans A Eriksson, MD, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D1443C00033
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quetiapine Fumarate Immediate Release
  Interventions: Drug: Quetiapine Fumarate
- 2 (Experimental): Quetiapine Fumarate Extended Release
  Interventions: Drug: Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate — Tablet, Oral, once daily
  Other Names: Seroquel IR
  Arms: 1
Drug: Quetiapine Fumarate — Tablet, Oral, once daily
  Other Names: Seroquel XR
  Arms: 2

SUMMARY:
This study will compare the tolerability of Quetiapine Fumarate immediate release formulation and Quetiapine Fumarate extended release formulation during initial dose escalation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Weight of at least 50 kg

Exclusion Criteria:

* A history or presence of neurological, hematological, psychiatric, gastrointestinal, hepatic, pulmonary, or renal disease or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Positive test results for alcohol or drugs of abuse
* Positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) 1 hour post dose at Day 1 | 1 hour after dose administration at the first dosing day (i.e. Day 1) of each period
Area under the VAS-time curve | Calculated daily from the 13 assessments for 5 days

SECONDARY OUTCOMES:
Pharmacodynamic relationship between maximum VAS and PK concentration | On last day of period (Day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Datto, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Datto C, Berggren L, Patel JB, Eriksson H. Self-reported sedation profile of immediate-release quetiapine fumarate compared with extended-release quetiapine fumarate during dose initiation: a randomized, double-blind, crossover study in healthy adult subjects. Clin Ther. 2009 Mar;31(3):492-502. doi: 10.1016/j.clinthera.2009.03.002. PMID 19393840